CLINICAL TRIAL: NCT03260101
Title: A Non-interventional, Long-term Follow-up of Subjects Who Completed ApoGraft-01 Study
Brief Title: Non-interventional, Long-term Follow-up of Subjects Who Completed ApoGraft-01 Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cellect Biotechnology (Industry)
Responsible Party: Sponsor
Other Study IDs: ApoGraft01 FU
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Acute Myelogenous Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Non Hodgkin Lymphoma (NHL); Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group, ApoGraft Follow up Study: Non-interventional, long-term follow-up study in subjects who received ApoGraft in study ApoGraft-01
  Interventions: Other: non intervational

INTERVENTIONS:
Other: non intervational — Subjects who completed ApoGraft-01 study (through 180 days post-transplantation) and have signed informed consent for this follow-up study will be eligible to enroll. Subject will attend 4 in-clinic visits, once every 6 months up to 2 years post transplantation, and will undergo the following evaluations: acute and chronic graft versus host disease (GvHD) assessments, survival status (overall, relapse-free), disease status (disease relapse/recurrence)
  Other Names: ApoGraft follow up

SUMMARY:
This is a non-interventional, long-term follow-up study in subjects who received ApoGraft in study ApoGraft-01. Up to 12 subjects who completed ApoGraft-01 study will be offered to participate in this follow-up study.

Subjects who completed ApoGraft-01 study and have signed informed consent for this follow-up study will be eligible to enroll. Subject will attend in-clinic visits up to 2 years post transplantation, and will undergo the following evaluations: acute and chronic graft versus host disease (GvHD) assessments, survival status (overall, relapse-free), disease status (disease relapse/recurrence), physical examination, safety laboratory and concomitant medication use.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who completed study ApoGraft-01 through 180 days (6 months) post-transplantation
2. Ability to comply with the requirements of the study.
3. Signed written informed consent

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 12 subjects who completed ApoGraft-01 study will be offered to participate in this follow-up study. Subjects must have had one of the Hemato-Oncology Diseases to enroll into ApoGraft-01:
  * Acute myelogenous leukemia (AML) & Acute lymphoblastic leukemia (ALL)
  * Non-Hodgkin's lymphoma (NHL)
  * Hodgkin's lymphoma (HL)
  * Intermediate, High or Very High risk Myelodysplastic syndrome (MDS)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2018-06-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, grade and stage of acute GvHD and chronic GvHD | 18 months
  GVHD will be assessed according to NIH criteria 2005; current and maximal score at each visit.

SECONDARY OUTCOMES:
Non-relapse-related mortality | 18 months
Proportion of subjects with disease relapse/recurrence | 18 months
Proportion of subjects with relapse free and overall survival | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No